CLINICAL TRIAL: NCT05201287
Title: A Pilot Study Evaluating the Safety and Clinical Effectiveness of Nucleus Pulposus Allograft for Supplementation of Nucleus Pulposus Tissue in Patients With Symptomatic Degenerated Discs
Brief Title: VIA Disc NP Pilot for Patients With Symptomatic Degenerated Discs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIVEX Biologics, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIA-2021-001
Record Dates: First submitted 2021-09-24; First posted 2022-01-21 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Disc Disease; Low Back Pain; Disc Degeneration
Keywords: low back pain; degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Up to 35 patients at 7 sites will receive treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VIA Disc Nucleus Pulposus Allograft (Experimental): A single dose, intradiscal injection of 100mg of VIA Disc NP mixed with 2ml sterile saline administered to the affected 1 or 2 levels, L1-S1.
  Interventions: Other: VIA Disc NP

INTERVENTIONS:
Other: VIA Disc NP — VIA Disc NP is processed from donated cadaveric disc tissue, lyophilized, and micronized to particles.
  Other Names: VIA Disc Nucleus Pulposus Allograft

SUMMARY:
VIA Disc NP is an allograft intended to supplement the nucleus pulposus tissue in degenerated intervertebral discs.

DETAILED DESCRIPTION:
The study will include adult subjects, ages 18 years or older, with symptomatic lumbar intervertebral disc degeneration that is not adequately resolved by non-surgical standard care. For the purpose of the primary analysis, subjects are considered enrolled in the study once they have signed the informed consent.

Each subject will receive one injection per level (max of 2 levels) and be evaluated for efficacy and safety during the up to 24 month observation period. The study is expected to be completed within 26 months, inclusive of enrollment and follow-up for all subjects.

Subjects will be evaluated at baseline and followed through up to 24 months to establish safety and efficacy of the treatment. The expected duration of subject participation from screening/enrollment through final follow-up is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

Eligibility for inclusion is evaluated on a site-specific basis based on each subject's medical, clinical, and radiographic presentation. In addition, for study consistency purposes, the MRI imaging will be submitted to Medical Metrics Imaging (MMI), a core lab, for independent review. MMI will review imaging of every subject to confirm radiographic inclusion criteria. The Medical Monitor will make the final determination for inclusion on all subjects based on review of the MRI relevant medical history and source documents.

1. Age 18 years or older;
2. Body mass index (BMI) < 35;
3. Documented diagnosis of moderate radiographic degeneration of up to 2 intervertebral discs from L1 to S1, with a suspected associated discogenic chronic low back pain;
4. Chronic LBP for ≥ 6 months;
5. Failed conservative care over the past 3 months of at least 2 conservative treatments including:

   1. oral pain medication [analgesics, steroids and/or non-steroidal anti-inflammatory drugs (NSAIDs)],
   2. structured physical therapy or exercise program prescribed by physical therapist, chiropractor, provider or physician specifically for the treatment of low back pain, and
   3. epidural steroid injections and/or facet injections/selective nerve blocks;
6. An MRI demonstrating:

   1. 1 to 2 vertebral level involvement L1-S1;
   2. Modified Pfirrmann Grade 3-7;
   3. No modic changes or if changes ≤ 2;
7. Oswestry Disability Index (ODI) score at time of evaluation of ≥ 40 and ≤ 80 points;
8. Low back pain of Baseline Numeric Rating Scale (NRS) score of ≥ 6 on the 11-point scale;
9. No signs or symptoms of current infection;
10. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study;
11. Be willing and able to comply with all study procedures and availability for the duration of the study with a life expectancy of > 2 years.

Exclusion Criteria:

1. Known allergies to Gentamicin, Vancomycin;
2. Contraindications to the proposed sedation/anesthetic protocol;
3. Radicular pain greater than back pain by history or evidence of radicular pain or neurological deficit within the past 6 months. Radicular pain is defined as nerve pain following a dermatomal distribution and that correlates with nerve compression on imaging. Somatic referred pain is allowed;
4. Any of the following conditions at the index level:

   1. Contained disc protrusion >5 mm or disc extrusion, or spondylolisthesis >5 mm (lysis and degenerative);
   2. Seronegative spondyloarthropathy;
   3. Symptomatic spinal stenosis (moderate to severe in degree);
   4. Chronic facet syndrome;
   5. Spondylodiscitis;
   6. Bilateral spondylolysis;
   7. Current or history of osteoporotic or tumor-related vertebral body compression fracture;
   8. Previous lumbar spine fusion surgery or disc arthroplasty;
5. History of sacroiliac (SI) joint pain/injections during the past 3 months or SI joint fusion within the past two years;
6. Received chemonucleolysis or percutaneous treatment of the affected disc prior to the study;
7. History of epidural steroid injections within 1 week prior to study treatment;
8. Received any lumbar intradiscal treatment injection or procedure (e.g., injection of methylene blue, dextrose, glucosamine, and chondroitin sulfate, or biacuplasty) and any nerve ablation procedures at the same or adjacent level (e.g., Basivertebral nerve ablation, dorsal ramus or sinovertebral nerve ablations). Discography and anaesthetic discography may be performed but must be done at least 2 weeks or more prior to the injection procedure;
9. Been a recipient of prior stem cell/progenitor cell therapy or other biological intervention (e.g., PRP) to repair the target intervertebral disc;
10. Severe motor deficit or cauda equina disorder based on investigator determination;
11. Diagnosis of any traumatic neurological disorders;
12. Severe diseases of any other major body system as judged by the investigator, including malignant diseases of any solid organ or any hematologic malignancy during the previous 5 years;
13. Demonstrate 3 or more Waddell's signs of Inorganic Behavior;
14. Any mental instability, bipolar disorders, post-traumatic stress disorder (PTSD) or uncontrolled anxiety/depression and/or require new or changed anti-depressants or anti-psychotic medications within 3 months of enrollment;
15. Compensated injuries or ongoing litigation regarding back pain/injury, or financial or other incentives to remain impaired;
16. If female and of child-bearing potential, are pregnant or breastfeeding or a plan to become pregnant or breastfeed in the first 12 months post-treatment;
17. Any medical condition that impairs follow-up (i.e., fibromyalgia, rheumatoid arthritis, chronic regional pain syndrome, reflex sympathetic dystrophy);
18. Evidence of substance abuse (including marijuana); Note: subjects using prescribed extended-release narcotics (e.g., fentanyl patch, MS Contin, oxycontin) within the 3 months prior to screening; subjects on long-acting opioids may be given option to wean off opiates before enrollment. Subjects on short-acting opiates (e.g., hydrocodone, oxycodone, tramadol, etc.) may be included and utilization monitored after the treatment;
19. Are currently receiving treatment with radiation, chemotherapy, immunosuppression, or chronic steroid therapy (prednisone, or its equivalent, use of up to 5 mg/qd is allowed, as well as inhalation steroids for asthma);
20. Active implantable devices, such as cardiac pacemakers, spinal cord stimulators, intrathecal pumps, etc.
21. Bilateral spondylolysis at any level;
22. Fracture of the spine, previous lumbar spine surgery or previous treatment of the target disc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Patient self-reporting of Functional Efficacy with no change in neurological status using the Oswestry Disability Index (ODI) | baseline to 3 months
  Evaluate the change from baseline in functional disability on the Oswestry Disability Index (ODI) measured from 0 (minimal disability) to 100 (maximal disability). The ODI is 10 categories of function to quantify disability due to low back pain.
Review of all Adverse Events for Safety of treatment and product | baseline to 6 months
  Evaluate the incidence of related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events from baseline through the final follow-up visit that are related to treatment and product.

SECONDARY OUTCOMES:
Patient self-reporting of Function | 3-6 months
  Owestry Disability Index (ODI) is measured 0 (minimal disability) to 100 (maximal disability). This index is comprised of ten categories of function to quantify disability due to low back pain. Functional responder analysis at 3 and 6 months measured as subjects meeting functional improvement of ≥ 10, 15 and 20 points in ODI scores.
Patient self-reporting of Pain | 3-6 months
  Changes in Numeric Rating Scale (NRS) scores. Eleven point pain scale used for patient self-reporting of back pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable). Analysis at 3 and 6 months measured as subjects meeting lower back pain NRS improvement of 50%.
Patient self-reporting of Pain in low back | 3-6 months
  Changes in Numeric Rating Scale (NRS) scores. Eleven-point pain scale used for patient to self-report level of back pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable). Analysis at 3 and 6 months measured as subjects meeting lower back pain NRS improvement of ≥30%.
Oswestry Disability Index (ODI) score change | baseline and 6 months
  Change from baseline in ODI scores at 6 months. Ten category index comprising of function to quantify due to low back pain. ODI is measured 0 (minimal disability) to 100 (maximal disability).
Numeric Rating Scale change | baseline, 3 and 6 months
  Changes from baseline in Numeric Rating Scale (NRS) score at 3 and 6 months. Eleven-point pain scale used for patient self-reporting of pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable).
Neurological status change | baseline to 6 months
  Change from baseline in motor function (graded 0 - no movement to 4 - active movement against resistance), reflexes (0 - absence to 4 - abnormal/hyperactive) and sensory status (graded normal or abnormal) based on physician's physical exam at 1, 3, and 6 months.
Return to work | baseline - 6 months
  Patient reported return to work - same or different capacity responses to employment questions will be assessed across time points and compared.
Magnetic Resonance Imaging (MRI) review to determine disc health changes | baseline-6 months
  Magnetic Resonance Imaging (MRI) taken at baseline compared to 6 months reviewing changes in treated disc levels (disc height, volume hydration of disc and Modified Pfirrman grade, T1rho relaxation, T2 relaxation for up to 10 subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Beall, MD, Principal Investigator — Clinical Radiology of Oklahoma
Locations (6):
- United States (6):
  - California Orthopedics and Spine, Larkspur, California
  - Source Health, Santa Monica, California
  - IPM Medical Group, Walnut Creek, California
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Virginia iSpine, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beall DP, Davis TT, Amirdelfan K, Naidu RK, DePalma MJ, Costandi S, Yoon ES, Fleming JW, Block JE, Mekhail N. Supplemental nucleus pulposus allograft in patients with lumbar discogenic pain: results of a prospective feasibility study. BMC Musculoskelet Disord. 2025 May 1;26(1):437. doi: 10.1186/s12891-025-08701-0. PMID 40312677